CLINICAL TRIAL: NCT01144286
Title: Multi-center, Randomized, Placebo-controlled, Parallel-group, Double-blinded Study to Compare the Therapeutic Efficacy, Safety, and Tolerability of 3 Single Vaginal Doses of Arasertaconazole Nitrate Pessaries in the Treatment of VVC
Brief Title: Arasertaconazole Nitrate Pessaries - Dose Finding Study for the Vulvovaginal Candidiasis (VVC) Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-090756-01; 2009-016655-21 (EudraCT Number)
Record Dates: First submitted 2010-06-09; First posted 2010-06-15 (Estimated); Results first posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-08

CONDITIONS: Vulvovaginal Candidiasis
Keywords: VVC; candidiasis; vaginal candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Candidiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator): placebo pessary, single dose
  Interventions: Drug: arasertaconazole nitrate
- Arasertaconazole nitrate 150 mg (Experimental): Arasertaconazole nitrate 150 mg pessary, single dose
  Interventions: Drug: arasertaconazole nitrate; Drug: placebo
- arasertaconazole nitrate 300 mg (Experimental): Arasertaconazole nitrate 300 mg pessary, single dose
  Interventions: Drug: arasertaconazole nitrate; Drug: placebo
- arasertaconazole 600 mg (Experimental): Arasertaconazole nitrate 600 mg pessary, single dose
  Interventions: Drug: arasertaconazole nitrate; Drug: placebo

INTERVENTIONS:
Drug: arasertaconazole nitrate — Arasertaconazole nitrate pessary, placebo pessary
Drug: placebo — placebo, single dose
  Arms: Arasertaconazole nitrate 150 mg; arasertaconazole 600 mg; arasertaconazole nitrate 300 mg

SUMMARY:
In order to find an optimal dose of arasertaconazole nitrate in the treatment of vulvovaginal candidiasis, a multicenter, randomized, double-blind, parallel, placebo-controlled study will be conducted to compare the therapeutic efficacy, safety and tolerability of three different doses of arasertaconazole nitrate (150 mg, 300 mg or 600 mg, pessaries).

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 to 65 years of age who have signed the informed consent.
* Not pregnant, not nursing.
* No indication of other vulvovaginitis or genital infections
* Positive 10% potassium hydroxide (KOH) preparation for budding yeast and/or pseudohyphae.
* Negative wet mount results for T. vaginalis and clue cells.
* Exclusion Criteria:
* Subjects with another vaginal or vulvar condition that would confound the interpretation of clinical response.
* Hypersensitivity to imidazole products administered topically.
* Any other medical condition which in the opinion of the investigator could interfere with study conduct.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ferrer Internacional S.A., Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were randomized to a treatment arm using an interactive web response system (IWRS). Placebo and study drug pessaries were dispensed as a kit, and all subjects were instructed in proper self-administration of the pessaries (at bedtime while lying down). Study initiation date was 15June2010 and completed on 15 Nov 2010.
Pre-assignment Details: After signed informed consent, VVC clinical signs and symptoms were assessed,(KOH) wet mounts and samples for mycological culture obtained.Baseline safety assessments, including pregnancy were performed. If all inclusion criteria and none of the exclusion criteria were met, the subject was randomized in the same day to one of the treatment groups.
Period: Overall Study
Arm/Group | Placebo | Arasertaconazole Nitrate 150 mg | Arasertaconazole Nitrate 300 mg | Arasertaconazole 600 mg
Started | 57 | 58 | 58 | 56
Completed | 57 | 58 | 58 | 56
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Arasertaconazole Nitrate 150 mg | Arasertaconazole Nitrate 300 mg | Arasertaconazole 600 mg | Total
Number analyzed (Participants) | 57 | 58 | 58 | 56 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 57 | 58 | 58 | 56 | 229
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.1 (7.74) | 32.8 (8.47) | 29.7 (7.58) | 31.8 (8.53) | 31.1 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 58 | 56 | 229
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Europe | 57 | 58 | 58 | 56 | 229

OUTCOME MEASURES:

1. Primary Outcome: Dose-response of Clinical and Mycological (Global) Therapeutic Response
Description: Global therapeutic response at day 26± 4 days ("TOC"- Test-of-Cure visit).Global therapeutic response is a composite endpoint using the clinical (signs and symptoms) and the mycological cures (microbiological culture), according to FDA guideline "Vulvovaginal Candidiasis -Developing Antimicrobial Drugs for Treatment".
Time Frame: day 26 ± 4 days
Population: The full analysis set (FAS) was the primary population for the analysis of all efficacy endpoints. The FAS was defined as all randomized subjects who received at least 1 dose of a study drug.Subjects in the FAS were analyzed according to randomized treatment group.
Measure: Number (95% Confidence Interval); unit: percentage of patients cured
Arm/Group | Placebo | Arasertaconazole Nitrate 150 mg | Arasertaconazole Nitrate 300 mg | Arasertaconazole 600 mg
Number analyzed (Participants) | 57 | 58 | 58 | 56
percentage of patients cured | 31.7 [18.08 to 48.09] | 48.7 [32.42 to 65.22] | 47.6 [32.00 to 63.58] | 53.8 [37.18 to 69.91]
Statistical Analysis 1: Comparison: Placebo vs Arasertaconazole Nitrate 150 mg vs Arasertaconazole Nitrate 300 mg vs Arasertaconazole 600 mg; Primary analysis is the dose response at TOC based on the global therapeutic cure. Dose response will be tested using a logistic regression using linear coefficient for the treatment effect(Wald chi-square). Assuming that the response rate is 80% for 600 mg, 75% for the 300 mg, 65% for 150 mg and 50% for the placebo group, a sample size of 45 subjects in each group will have 90% power to detect a linear dose response using a 0.05 two-sided test of trend based on the logistic model; Test type: Superiority or Other; p = 0.0630, Regression, Logistic — Significance level was set to α of 0.05 if the primary endpoint was significant, hierarchical testing was to be performed on the primary endpoint (each active dose X placebo). No other adjustment was made for testing multiple secondary outcomes; response rate (%) = 80

2. Secondary Outcome: Dose-response of Clinical and Mycological (Global)Therapeutic Response
Description: Global therapeutic response at day 8± 2 days. Safety and tolerability.
Time Frame: Day 8 ± 2 days
Population: Dose response tested using logistic regression-linear coefficient for treatment effect.Assuming response rate 80% for 600 mg, 75% for 300 mg, 65% for 150 mg and 50% for the placebo group, sample size of 45 subjects in each group have 90% power to detect linear dose response with 0.05 two-sided test of trend based on the logistic model.
Measure: Number (95% Confidence Interval); unit: percentage of cured participants
Arm/Group | Placebo | Arasertaconazole Nitrate 150 mg | Arasertaconazole Nitrate 300 mg | Arasertaconazole 600 mg
Number analyzed (Participants) | 57 | 58 | 58 | 56
percentage of cured participants | 15.6 [6.49 to 29.46] | 34.2 [19.63 to 51.35] | 46.3 [30.66 to 62.58] | 61.0 [44.50 to 75.80]

ADVERSE EVENTS:
Time Frame: Study Initiation Date: 15 June 2010 Study Completion Date: 15 November 2010
Arm/Group | Placebo | Arasertaconazole Nitrate 150 mg | Arasertaconazole Nitrate 300 mg | Arasertaconazole 600 mg
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/58 | 0/58 | 0/56
Other Adverse Events (participants affected / at risk) | 6/57 | 9/58 | 13/58 | 13/56
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | Arasertaconazole Nitrate 150 mg (N=58) | Arasertaconazole Nitrate 300 mg (N=58) | Arasertaconazole 600 mg (N=56)
tonsilitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — moderate, not related,recovered
Chamydial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild, not related, recovering
heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild, not related, recovered
headache (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) — mild, not related, recovered
vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — mild, possible related, recovered
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — mild, not related, recovered
abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — mild, possible related, recovered
vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — mild, not related, recovered
nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — mild, not related, recovered
respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — mild, not related, recovered
rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — mild, not related, recovered
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — moderate, unlikely, recovered
arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) — mild, unlikely, recovered
vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — mild, unlikely, recovered
bloody discharge (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — mild, possible related, recovered
influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — mild-moderate, not related, recovered
electrocardiogram TWave decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — moderate, not assessable, recovered
pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — There were 2 pregnancy cases. Patient exposed to 600 mg Arasertaconazole delivered healthy boy at 38th week gestation. Investigator last report received patient exposed to 300 mg Arasertaconazole: Ultrasound at 20th week of gestation was normal.
vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — severe, probable related, recovered
dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — moderate, not related, recovered
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild, not related, recovered
vaginitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild, not related, recovered
blood bilirrubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild, not related, not recovered
migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild, not related, recovered
urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — moderate, possible related, recovered
pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — moderate, not related, recovered
uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — mild, possible related, recovered
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild, not related, recovered
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild, not related, recovered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review publications and/or presentations (results communications) prior to public release and communications regarding trial results for a period that is 60 days from the time submitted to the sponsor for review. The sponsor may require changes to the publication and /or presentation regarding its content or the time of release.